CLINICAL TRIAL: NCT06794359
Title: Minimally Invasive Coronary Artery Bypass Surgery: Prospective and Randomized Study to Validate the Minimally Invasive Approach Through Left Anterior Mini Thoracotomy in Patients With Milti Vessel Coronary Disease
Brief Title: Minimally Invasive Coronary Artery Bypass Surgery in Patients With Multi Vessel Coronary Disease
Acronym: MINICABG
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Medtronic (Industry); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Luís Alberto Oliveira Dallan, Cardiovacular Surgeon, Director of the Coronary Artery Disease Division at the HC Heart Institute - FMUSP, Associated Professor FMUSP, PhDr in health sciences, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE 54175921.8.0000.0068; 2021/11947-5 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2024-10-14; First posted 2025-01-27 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Coronary Arterial Disease (CAD); Coronary Artery Bypass
Keywords: CABG; MICS CABG; CAD
MeSH Terms: interventions — Coronary Artery Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minimally Invasive Coronary Artery Bypass (Experimental): Experimental: Minimally Invasive Coronary Artery Bypass will be performed in a through left anterior mini thoracotomy. Complete revascularization must be performed in all previous determined coronary targets.
  Interventions: Procedure: Minimally Invasive Coronary Artery Bypass Grafting
- Conventional Coronary Artery Bypass Grafting (Active Comparator): Conventional Coronary Artery Bypass Grafting will be performed in a classic manner, through total sternotomy. Complete revascularization must be performed in all previous determined coronary targets.
  Interventions: Procedure: Coronary artery bypass surgery

INTERVENTIONS:
Procedure: Minimally Invasive Coronary Artery Bypass Grafting — Minimally Invasive Coronary Artery Bypass Grafting will be accomplished by complete revascularization of all previous defined coronary targets through left anterior thoracotomy. On or off pump approach will be determined by the surgeon. For on pump cases, femoral canulation will be performed and aortic cross clamp will be used. Off Pump cases will be performed using Medtronic Octopus and Starfish NS. Intra operative Transit time flow measurement will be performed in all cases.
  Arms: Minimally Invasive Coronary Artery Bypass
Procedure: Coronary artery bypass surgery — Procedure: Conventional Coronary Artery Bypass Grafting will be accomplished by complete revascularization of all previous defined coronary targets through classical total sternotomy. On or off pump approach will be determined by the surgeon. Intra operative Transit time flow measurement will be performed in all cases.
  Arms: Conventional Coronary Artery Bypass Grafting

SUMMARY:
The objective of this study is to evaluate the safety and feasibility of Minimally Invasive Coronary Artery Bypass surgery in selected patients ,with multi vessel coronary disease.

This trial is designed to be a pilot study that will gather comparative information on the clinical performance of the minimally invasive treatment, evaluated by the composite measure of all-cause death, myocardial infarction, stroke, or unplanned repeat revascularization - in hospital, 30-day and 6 months.

DETAILED DESCRIPTION:
Minimally invasive surgery has been a breakthrough in medicine, especially in more developed countries. It represents an evolution of current techniques associated with new technologic devices, that allow a safe and effective procedure associated to an aesthetic benefit.

Invasive treatment of coronary artery disease has been on a plateau lately. Percutaneous treatment that emerged as a promise to replace surgical methods, has already shown its limitations, even with the use of drug-eluting stents. Traditional CABG (coronary artery bypass grafting surgery), which has been considered the gold standard, has been criticized for its high degree of invasiveness.

Based on this precept, interest has emerged in creating a surgical approach that causes less trauma. Surgical access using minimally invasive incisions are gaining space and have shown less postoperative pain, shorter hospital stays, earlier mobilization and functional recovery, in addition to reducing the costs of the procedure.

Cardiac surgery has some challenges that are beyond other specialties. The heart is a vital organ with intrinsic chronotropism that lies inside a rigid rib cage.

Specifically, in coronary artery bypass graft surgery (CABG), the thin caliber of the coronaries and their distribution throughout the cardiac territories creates even a greater challenge. However, new surgical techniques associated with new devices, demonstrated the viability of complete revascularization through a limited access incision.

In an attempt to minimize surgical trauma and the morbidities caused by conventional median sternotomy and the use of On Pump surgery, some alternatives have emerged with promising results.

Among those efforts, we can highlight the beginning of the coronary artery grafting surgery without the use of cardiopulmonary bypass (Off Pump CABG), followed by hybrid revascularization, minimally invasive surgery by lateral thoracotomy under direct vision, partially assisted robot surgery and fully endoscopic surgery with using robots.

Currently, minimally invasive surgery though mini lateral thoracotomy is the most common technique used. Initially it was used only for the treatment of the left anterior descending artery (LAD), but technology advances and surgical improvement allowed complete revascularization under direct vision. Surgery can be performed with or without the aid of cardiopulmonary bypass (CPB), treatment individualization is necessecary for every case.

This is a pilot study to evaluate the safety and feasibility of Minimally Invasive Coronary Artery Bypass surgery in selected patients ,with multi vessel coronary disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-years-old or older
* Isolated myocardial revascularization procedure
* Double or Triple-vessel disease with proximal or mid LAD disease with angiographic diameter stenosis > 70% by visual analysis in all territories, requiring myocardial revascularization OR proximal LAD disease with angiographic diameter stenosis 50-70% by visual analysis in any territory but with invasive or non-invasive evidence of flow-limiting stenosis in all three territories, requiring myocardial revascularization
* Total SYNTAX score > 22 or low Syntax score unsuitable for PCI
* Clinical and anatomic eligibility for both Minimally invasive and Conventional CABG surgery as agreed to by surgical team.
* Silent ischemia, stable angina, unstable angina or recent MI

  - If recent MI, cardiac biomarkers must have returned to normal prior to randomization
* Ability to sign informed consent and comply with all study procedures

Exclusion Criteria:

* Reoperation
* Need for any concomitant cardiac surgery other than CABG (e.g. valve surgery, aortic repair, etc.), or intent that if the patient randomizes to surgery, any cardiac surgical procedure other than isolated CABG will be performed
* Left ventricle disfunction (EF<40%)
* Chronic Pulmonary obstructive disease
* Renal failure disease
* Emergency surgery
* Obesity
* Sternum anatomic defects including pectus excavatum
* Peripheral vascular disease
* Ascending aorta severe calcification
* Non cardiac co-morbidities with life expectancy less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility and safety of proposed revascularization through minimally invasive approach | Clinical follow-up intra hospitalar, 30-day and 6 months
  This is a pilot study that wants to evaluate the feasibility of performing complete CABG through minimamlly invasive access, in patients with multi vessel disease (2 or more diseased coronaries), without compromising safety measured by major adverse events (death, myocardial infarction, stroke, or unplanned revascularization)

SECONDARY OUTCOMES:
Intraoperative conversion rate | Intraoperative measure
  Conversion rate
  * Off Pump to On Pump surgery (regardless of mini thoracotomy or conventional sternotomy)
  * mini thoracotomy to conventional sternotomy
Complete revascularization rate | Intraoperative measure
  Surgical team will define preoperatively the number of coronaries to be grafted. After the surgical procedure is completed, the number of performed grafts will be compared to the initial plan. Incomplete revascularization will be considered if the number of grafts performed is lower than the predicted. This is important to measure feasibility
Postoperative bleeding volume | First 48 hours post-surgery
  Postoperative bleeding volume will be measured in the first 48 hours after surgery. It will also be correlated to pre and postoperative hematocrit values. Blood flow transfusions during surgery and 24 hours after surgery will be measured.
Surgery duration | Intraoperative measure
  Surgery duration (hours) will be timed from the skin incision until skin dressing is finished.
Length of orotracheal intubation | From oral intubation until extubation
  Orotracheal intubation will be measured in hours from the oral intubation to extubation
Length of ICU and hospital stay | From ICU admission to discharge
  Length of ICU and hospital stay (days) will be timed from patient's entry on the sector until medical discharge is determined by intensive care and/or cardiology teams.
Intra operative graft evaluation | This is a specific assessment carried out during the surgical procedure (intraoperative).
  Intra operative time flow measurement (TTFM) allows measuring the graft flow using the MedStim devices.
  Three variables are analyzed: Graft flow, pulsatility index and diastolic flow percentage.
  Normal flow measures are expected to be over 15ml/min, pulsatility index is expected to be lower than 5 and diastolic flow percentage is expected to be over 50%.
  This is an important and specific assessment carried out exclusively during the surgical procedure.
  If the values found in the data differ from the data considered normal (shown above), reevaluation of the graft through exploration of the anastomosis should be considered.
  This values will be compared in the group of patients operated through regular sternotomy and those operated through left mini thoracotomy. If statistical differences are found it could suggest that the quality of the anastomosis colud differ between techniques
Postoperative myocardial infarction | Within 48 hours following surgery
  Periprocedural myocardial infarction (type 5 MI) will be defined according to the Fourth Universal Definition of Myocardial Infarction (UDMI-4, 2018) as an elevation of cardiac troponin values greater than 10 times the upper reference limit (URL) in patients with normal baseline levels, accompanied by at least one of the following objective indicators of myocardial ischemia: New pathological Q waves on electrocardiogram; new left bundle branch block; new regional motion abnormalities on echocardiography; angiography evidence of new occlusion of a native coronary artery or bypass graft.
  To enhance methodological rigor and allow comparison with contemporary clinical trials, the periprocedural MI definition proposed by the Academic Research Consortium-2 (ARC-2) will also be adopted as a secondary criterion, which includes: Troponin elevation >70× URL, or CK-MB elevation >10× URL, in association with hemodynamic instability, need for circulatory support.
Surgical Mortality | 30 days postoperatively
  Operative mortality and is defined as:
  1. all deaths, regardless of cause, occurring within 30 days from the procedure (including patients transferred to other care facilities);
  2. all deaths, regardless of cause, occurring after discharge from the hospital, but before the end of the 30th postoperative day (except for traumatic / external causes)
Wound infection | From the date of surgery through 30 days postoperatively.
  Wound infection will be defined by the presence of phlogistic signs at the incision, associated to the presence of purulent secretion and laboratorial exams.
Post operatative atrial fibrillation | Immediate postoperative: from the day of surgery to postoperative day 7. • Early late postoperative: from postoperative day 8 to day 30. • Late outpatient assessment: between 30 days and 6 months post-surgery.
  Postoperative atrial fibrillation (AF) will be defined as any new-onset episode requiring medical treatment, excluding patients with a prior or chronic history atrial fibrillation. Time Frame: AF assessment will be assessed at three time points:
  * Immediate postoperative: from the day of surgery to postoperative day 7.
  * Early late postoperative: from postoperative day 8 to day 30.
  * Late outpatient assessment: between 30 days and 6 months post-surgery.
Neurological events | Stroke related to surgery will be acessed in phases: • Immediate postoperative: from the day of surgery to postoperative day 7. • Early late postoperative: from postoperative day 8 to day 30. • Late outpatient assessment: between 30 days and 6 months po
  Procedure related stroke will be defined as a new neurological deficit lasting more than 72 hours, confirmed by neurological examination and brain imaging (computed tomography and/or magnetic resonance), with interpretation by a neurologist. Stroke assessment will be performed at threetime points:
  * Immediate postoperative: from the day of surgery to postoperative day 7.
  * Early late postoperative: from postoperative day 8 to day 30.
  * Late outpatient assessment: between 30 days and 6 months post-surgery.
Quality of Life Assessed by EQ-5D-5L | Within 6 Months After Surgery
  Postoperative quality of life will be assessed using the EuroQol EQ-5D-5L questionnaire, administered by telephone within 6 months after surgery.
Safety Assessed by Incidence of Major Adverse Cardiovascular and Cerebral Events (MACCE) Postoperatively | At 30 days and 6 months following hospital discharge
  Left anterior minithoracotomy surgery will be considered safe if the patient's postoperative recovery occurs with similar incidence of of major cardiac or cerebral events, as compared to the classical sternotomy (considered the gold standard procedure).
  Safety will be measured by major cariovascular and cerebral events, that include:
  * Cause of death (cardiac vs. non-cardiac);
  * Myocardial infarction type
  * stroke type and severity.
  All this variables mentioned are described with details on its respectives outcomes measures

CONTACTS AND LOCATIONS:
Overall Officials: Luis Roberto Palma Dallan, MD, Study Director — INCOR - Heart Institute from the University of Sao Paulo; Luis Alberto Oliveira Dallan, MD PhD, Principal Investigator — INCOR - Heart Institute from the University of Sao Paulo
Locations (1):
- INCOR - Heart Institute from the University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Necessary data will be shared uppon request, preserving patient's identification. (information that underlie results in a publication)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: This data will be avalilable 6 months after publication.
Access Criteria: Journal Editor whrere the paper will be accepted for publication. Other researchers who might want to cooperate on future reseaches.

REFERENCES:
- [Derived] Palma Dallan LR, Ferreira Lisboa LA, Oliveira Dallan LA, Asdrubal Vilca Mejia O, Neves Filho AF, Doenst T, Babliak O, Orellana Sampedro GA, Jatene FB. Minimally invasive coronary artery bypass grafting (MINI-CABG): Protocol for a pilot randomized controlled trial comparing minimally invasive versus conventional coronary surgery. PLoS One. 2025 Dec 29;20(12):e0337829. doi: 10.1371/journal.pone.0337829. eCollection 2025. PMID 41460930